CLINICAL TRIAL: NCT04833023
Title: HALO Trial: Haloperidol vs Olanzapine in Hyperactive Delirium in Palliative Care Patients; A Multi-Centre, Randomised-Controlled Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Mervyn Koh Yong Hwang, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PalC-RG-20/P001
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Haloperidol; Advanced Cancer; Hyperactive Delirium; Olanzapine; End-stage Organ Disease
MeSH Terms: interventions — Haloperidol; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study statistician will be blinded to the treatment allocation and outcome assessments (for example, Richmond Agitation and Sedation Scale).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Haloperidol Arm (Active Comparator): Haldol 2mg/ml oral solution
  Interventions: Drug: Haldol 2mg/ml oral solution
- Olanzapine Arm (Active Comparator): Olanzapine Actavis 5mg orodispersible tablet
  Interventions: Drug: Olanzapine Actavis 5mg orodispersible tablet

INTERVENTIONS:
Drug: Haldol 2mg/ml oral solution — Starting dose: 1mg
  Maximum Dose within 24 hours: 6mg
  Doses can be escalated every 2 hourly to the maximum doses allowed within 24 hours. If maximum dose of Haloperidol has been reached for the day (within 24 hours), rescue dose of Midazolam 2mg can be used (2mg Q2H PRN).
  Arms: Haloperidol Arm
Drug: Olanzapine Actavis 5mg orodispersible tablet — Starting dose: 2.5mg
  Maximum Dose within 24 hours: 15mg
  Doses can be escalated every 2 hourly to the maximum doses allowed within 24 hours. If maximum dose of Olanzapine has been reached for the day (within 24 hours), rescue dose of Midazolam 2mg can be used (2mg Q2H PRN).
  Arms: Olanzapine Arm

SUMMARY:
1. Background and Clinical Need:

   Delirium is common at the end of life and is challenging to control. There is a clinical need to study the benefits of commonly used drugs like Haloperidol and Olanzapine in the management of hyperactive delirium in advanced cancer or end-stage organ disease patients in a scientifically robust manner.
2. Aims/Hypotheses:

   The investigators aim to study the effectiveness of Haloperidol compared with Olanzapine in the management of hyperactive delirium in advanced cancer or end-stage organ disease patients receiving palliative care. The investigators hypothesise that Olanzapine is as effective as Haloperidol in the control of hyperactive delirium.
3. Methods:

   The investigators will conduct a pragmatic, multi-centre, (hospital, inpatient hospice, community hospital) open-label randomised-controlled trial comparing the use of Haloperidol versus Olanzapine in advanced cancer or end-stage organ disease patients with hyperactive delirium.

   The primary outcome is the change in Richmond Agitation and Sedation Scale (RASS) scores among patients in each treatment group at 8 hours post-drug administration.

   The secondary outcome is the control of hyperactive delirium at 24, 48 and 72 hours using either Haloperidol or Olanzapine.

   The mean doses of Haloperidol and Olanzapine used as well as the volume of rescue Midazolam required as well as side-effects of the study medications, survival after enrolment into study will also be studied.
4. Significance to palliative care The results of this study will advance the knowledge of delirium management worldwide with regards to the efficacy of Haloperidol and Olanzapine in managing hyperactive delirium in patients with advanced cancer or end-stage organ disease.

Haloperidol is used traditionally in palliative care for managing delirium. However, as a conventional anti-psychotic, it does cause extra-pyramidal side-effects. Olanzapine, a newer atypical anti-psychotic with a more favourable side-effect profile is being used increasingly in the control of delirium. These 2 commonly used drugs have never been compared head to head in a randomised-controlled, multi-centre study.

DETAILED DESCRIPTION:
(A) Background & Clinical Need

Delirium is commonly encountered in palliative care with a prevalence of between 26-74% and rising to as high as 88% nearer the end of life (2). It negatively impacts patient care and leads to greater morbidity and mortality (3). There are 3 sub-types of delirium - hyperactive, mixed and hypoactive (4) with majority of well-designed studies in palliative care focusing on the management of delirium as a whole (5). However, recently published literature suggests that these delirium subtypes appear to have different trajectories and are also generally treated differently (6).

Overall, the management of delirium in palliative care remains controversial. Agar had shown in a randomised controlled trial that supportive care may be superior to the use of anti-psychotics, even though the patients in Agar's study were only 'mildly' delirious and the overall doses of anti-psychotics used was lower than compared to common practice (9). Other studies have shown the benefits of anti-psychotics like haloperidol, olanzapine and aripiprazole in the management of delirium (10,11).

Hui et al was the only study which looked at the management of hyperactive delirium in the palliative care setting (7). Patients with hyperactive delirium exhibit restlessness, agitation and even aggression towards their loved ones and to healthcare providers caring for them (8).

To date, there have not been any multi-centre, randomised-controlled trial which has addressed the effectiveness of oral Haloperidol vs Olanzapine in the management of hyperactive delirium in the palliative care setting.

(B) Specific Aims

The investigators aim to study the effectiveness of Olanzapine vs Haloperidol in the management of hyperactive delirium in patients with advanced cancer or end-stage organ disease in 3 different settings.

The primary outcome is the change in Richmond Agitation and Sedation Scale (RASS) scores among patients in each treatment group at 8 hours after the administration of Haloperidol or Olanzapine as measured using the Richmond Agitation and Sedation Scale (RASS).

The secondary outcome is the change in Richmond Agitation and Sedation Scale (RASS) score at 24, 48 and 72 hours with the use of either Haloperidol or Olanzapine required.

The mean doses of Haloperidol and Olanzapine used as well as the doses of rescue Midazolam required as well as side-effects of the study medications, survival after enrolment into study will also be studied.

(C) Methods

Study Design

The investigators aim to conduct a multi-centre, randomised-controlled, open-label trial (Acute Hospital Palliative Care Unit, Palliative Care Unit in Community Hospital and Inpatient Hospice) comparing the use of haloperidol vs olanzapine in a 1:1 ratio in advanced cancer or end-stage organ disease patients with hyperactive delirium. Patients will be followed up for 3 days (72 hours) with regards to the response to study medications as well as other factors and outcomes as described below. Mortality data will also be collected.

The study will be conducted in 3 different Palliative Care Centres in Singapore - 1. Tan Tock Seng Hospital Acute Palliative Care Unit, 2. Palliative Care Unit in St Andrews' Community Hospital and 3. Dover Park Hospice. This is to increase the pragmatic applicability and external validity in this study to different palliative care units in Singapore and internationally.

Informed consent will be taken from the patient's legal representative according to the HBR Act as the patients recruited will be delirious and therefore will not able to provide informed consent adequately.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer or end-stage organ disease
2. Age ≥ 21 years old
3. Fulfil All Three Diagnosis of Delirium:

   * Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria for delirium
   * Memorial Delirium Assessment Scale (MDAS)©1996 >/= 13
   * Richmond Agitation-Sedation Scale (RASS) Score +1 to +3
4. Able to consume medications orally
5. Prognosis > 48 hrs (Clinician Estimate)

Exclusion Criteria:

1. Parkinson's Disease or Vascular Parkinsonism
2. Patient with dementia
3. Chronic Schizophrenia on regular Anti-psychotic medications
4. Taking any regular Benzodiazepines* or any Anti-psychotic** medications
5. Known allergy to Haloperidol or Olanzapine
6. History of Substance Abuse
7. Known Prolonged corrected QT interval (QTc) Syndrome (In Patient's Medical History)
8. Prognosis < 48 hours (Clinician's Estimate)
9. Unable to consume oral medications
10. Richmond Agitation and Sedation Scale (RASS) Score +4 (Too agitated and will require Parenteral Anti-psychotics and/or Benzodiazepines)
11. Pregnancy * e.g. Lorazepam, Alprazolam, Clonazepam, Midazolam **e.g. Haloperidol, Risperidone, Quetiapine, Olanzapine

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Richmond Agitation and Sedation Scale (RASS) score | 8 hours
  The change in Richmond Agitation and Sedation Scale (RASS) score 8 hours after administration of either Haloperidol and Olanzapine. Minimum value is -5 which represents that the patient is in hypoactive delirium and is unarousable and maximum value is +4 with the higher score representing that the patient is in hyperactive delirium and is combative. The aim of the study is to reduce the hyperactive delirium to a score of 0 which represents patient is alert and calm.

SECONDARY OUTCOMES:
Comparing Patient and Family's concurrence on state of delirium with of the Diagnosis of Delirium from Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria for delirium. | 72 hours
  There have not been any studies that looked at interviewing patients who are delirious about their acknowledgement and concurrence of their state of delirium. The investigators aim to interview patients by asking the patient 'Did you feel confused' and caregivers similarly by asking 'Do you feel that your loved one is Confused' as shown as an example below and compare this to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria for delirium.
  Please ask the Patient the following question "Do you feel that you are confused?"
  1. Yes/Sometimes
  2. No
  3. Not Sure/ Unable to answer Please ask the Family member or Caregiver the following question "Do you think the patient is confused?"
  1) Yes/Sometimes 2) No 3) Not sure/ Unable to answer
Mean dose used of Haloperidol and Olanzapine | 72 hours
  Mean doses of Haloperidol and Olanzapine used at 8hours / D1 / D2 / D3 from the first time-point that the study medication is administered to the patients
Mean Time to control of Hyperactive Delirium | 72 hours
  Mean Time to control of Hyperactive Delirium
Rescue Psychotropic (Mean Doses): Midazolam | 72 hours
  Rescue Psychotropic (Mean Doses): Midazolam
Side-effects of Study Medications | 72 hours
  Side-effects of Study Medications
Survival time in days | 72 hours
  Survival time in days
Edmonton Symptom Assessment Score revised (ESAS-r) | 1 hour
  Edmonton Symptom Assessment Score revised (ESAS-r) - At the point of recruitment
  Minimum value for the scale is 0 and maximum value for the scale is 10 with the higher value representing worse outcome.
Memorial Delirium Assessment Score (MDAS) | 72 hours
  Memorial Delirium Assessment Score (MDAS) - At the point of recruitment and after 72 hours
  It is a scale comprising of 10 items with scores of 0-3 for each question. Add up the score for all 10 questions and scores with more than or equal to 13 point indicates delirium.
Richmond Agitation and Sedation Scale (RASS) score | 72 hours
  Richmond Agitation and Sedation Scale (RASS) score: 8hours / 24hours (Day 1) / 48 hours (Day 2) / 72 hours (Day 3)
  Minimum value is -5 which represents that the patient is in hypoactive delirium and is unarousable and maximum value is +4 with the higher score representing that the patient is in hyperactive delirium and is combative. The aim of the study is to reduce the hyperactive delirium to a score of 0 which represents patient is alert and calm.
Caregiver and Nurses Perception on the control of hyperactive delirium | 72 hours
  Caregiver and Nurses Perception on the control of hyperactive delirium (5-point Likert Scale). Kindly refer to the example of the question below.
  The patient is less agitated as compared to 72 hours ago? (Clinician/Nurse):
  1. - Strongly Disagree
  2. - Disagree
  3. - Neutral
  4. - Agree
  5. - Strongly Agree
  The patient is less agitated as compared to 72 hours ago? (Family/Caregiver):
  1. - Strongly Disagree
  2. - Disagree
  3. - Neutral
  4. - Agree
  5. - Strongly Agree

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Koh, Principal Investigator — Tan Tock Seng Hospital
Locations (3):
- Singapore (3):
  - Tan Tock Seng Hospital, Singapore
  - Dover Park Hospice, Singapore
  - St. Andrew's Community Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data available to other researchers.

REFERENCES:
- [Background] Hosie A, Davidson PM, Agar M, Sanderson CR, Phillips J. Delirium prevalence, incidence, and implications for screening in specialist palliative care inpatient settings: a systematic review. Palliat Med. 2013 Jun;27(6):486-98. doi: 10.1177/0269216312457214. Epub 2012 Sep 17. PMID 22988044
- [Background] Watt CL, Momoli F, Ansari MT, Sikora L, Bush SH, Hosie A, Kabir M, Rosenberg E, Kanji S, Lawlor PG. The incidence and prevalence of delirium across palliative care settings: A systematic review. Palliat Med. 2019 Sep;33(8):865-877. doi: 10.1177/0269216319854944. Epub 2019 Jun 11. PMID 31184538
- [Background] Hui D. Delirium in the palliative care setting: "Sorting" out the confusion. Palliat Med. 2019 Sep;33(8):863-864. doi: 10.1177/0269216319861896. No abstract available. PMID 31395002
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Skelton L, Guo P. Evaluating the effects of the pharmacological and nonpharmacological interventions to manage delirium symptoms in palliative care patients: systematic review. Curr Opin Support Palliat Care. 2019 Dec;13(4):384-391. doi: 10.1097/SPC.0000000000000458. PMID 31490322
- [Background] Zipser CM, Knoepfel S, Hayoz P, Schubert M, Ernst J, von Kanel R, Boettger S. Clinical management of delirium: The response depends on the subtypes. An observational cohort study in 602 patients. Palliat Support Care. 2020 Feb;18(1):4-11. doi: 10.1017/S1478951519000609. PMID 31506133
- [Background] Hui D, Frisbee-Hume S, Wilson A, Dibaj SS, Nguyen T, De La Cruz M, Walker P, Zhukovsky DS, Delgado-Guay M, Vidal M, Epner D, Reddy A, Tanco K, Williams J, Hall S, Liu D, Hess K, Amin S, Breitbart W, Bruera E. Effect of Lorazepam With Haloperidol vs Haloperidol Alone on Agitated Delirium in Patients With Advanced Cancer Receiving Palliative Care: A Randomized Clinical Trial. JAMA. 2017 Sep 19;318(11):1047-1056. doi: 10.1001/jama.2017.11468. PMID 28975307
- [Background] Breitbart W, Alici Y. Agitation and delirium at the end of life: "We couldn't manage him". JAMA. 2008 Dec 24;300(24):2898-910, E1. doi: 10.1001/jama.2008.885. PMID 19109118
- [Background] Agar MR, Lawlor PG, Quinn S, Draper B, Caplan GA, Rowett D, Sanderson C, Hardy J, Le B, Eckermann S, McCaffrey N, Devilee L, Fazekas B, Hill M, Currow DC. Efficacy of Oral Risperidone, Haloperidol, or Placebo for Symptoms of Delirium Among Patients in Palliative Care: A Randomized Clinical Trial. JAMA Intern Med. 2017 Jan 1;177(1):34-42. doi: 10.1001/jamainternmed.2016.7491. PMID 27918778
- [Background] Boettger S, Friedlander M, Breitbart W, Passik S. Aripiprazole and haloperidol in the treatment of delirium. Aust N Z J Psychiatry. 2011 Jun;45(6):477-82. doi: 10.3109/00048674.2011.543411. PMID 21563866
- [Background] Lin CJ, Sun FJ, Fang CK. An open trial comparing haloperidol with olanzapine for the treatment of delirium in palliative and hospice center cancer patients. J Internal Med Taiwan 2008; 19:346-354.
- [Background] Bush SH, Grassau PA, Yarmo MN, Zhang T, Zinkie SJ, Pereira JL. The Richmond Agitation-Sedation Scale modified for palliative care inpatients (RASS-PAL): a pilot study exploring validity and feasibility in clinical practice. BMC Palliat Care. 2014 Mar 31;13(1):17. doi: 10.1186/1472-684X-13-17. PMID 24684942